CLINICAL TRIAL: NCT02164812
Title: A Study to Determine the Concentration-Electrocardiographic Effects of Efavirenz in Healthy Subjects Enriched for CYP2B6 Polymorphisms
Brief Title: Study to Determine the Effect of Efavirenz on the ECG QTcF Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AI266-959
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Moxifloxacin; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moxifloxacin, Placebo, Efavirenz (Experimental): Moxifloxacin, Placebo, Efavirenz single dose as specified
  Interventions: Drug: Moxifloxacin; Drug: Placebo; Drug: Efavirenz

INTERVENTIONS:
Drug: Moxifloxacin
  Other Names: Avelox®
Drug: Placebo
Drug: Efavirenz
  Other Names: Sustiva®; BMS-561525

SUMMARY:
The purpose of this study is to determine whether multiple doses of Efavirenz has an effect on the QTc interval (corrected by Fridericia) in CYP2B6 *1/*6 and *6/*6 healthy subjects.

DETAILED DESCRIPTION:
CYP = Cytochrome p-450

Primary Purpose: Other: This is a Phase 1 clinical pharmacology thorough QT study being conducted as a post marketing requirement

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy volunteers, ages 18 to 49 years old
* BMI 18 to 32 kg/m2
* Women must not be pregnant or breastfeeding

Exclusion Criteria:

* A personal history of clinically relevant cardiac disease, symptomatic or asymptomatic arrhythmias, presyncope or syncopal episodes, or additional risk factors for torsades de pointes (eg, heart failure)
* History of hypokalemia, personal history or family history of prolonged QT interval, or family history of sudden cardiac death at a young age
* Any of the following on 12-lead electrocardiogram (ECG) prior to study drug administration: PR ≥210 msec, QRS ≥120 msec, QT ≥500 msec, QTcF ≥450 msec, HR <45 bpm
* Second or third degree heart block prior to study drug
* Positive urine screen for drugs of abuse
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or Human Immunodeficiency Virus (HIV)-1, -2 antibody
* Any of the following lab results outside of the ranges specified below prior to dosing: Alanine aminotransferase (ALT) >upper limit of normal (ULN), aspartate aminotransferase (AST) >ULN, Total bilirubin >ULN, Direct bilirubin >ULN, Creatinine >ULN, Serum potassium <lower limit of normal (LLN), Serum magnesium <LLN
* History of allergy to Moxifloxacin, Efavirenz or related compounds

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Difference from placebo of Efavirenz (EFV) in change from period-specific baseline in the QT interval corrected for heart rate (HR) via Fridericia's method (QTcF) at postdose extraction times (ΔΔQTcF) | Days 1, 2, 5, 6, 19 and 20
  QTcF = QT corrected for Fridericia's formula

SECONDARY OUTCOMES:
Difference from placebo of EFV in change from period-specific baseline in other ECG parameters: HR, PR, QRS, and uncorrected QT following 14 days of dosing | Days 1, 5 and 19
  ECG = Electrocardiogram
Difference from placebo of Moxifloxacin in change from period-specific baseline in QTcF (ΔΔQTcF) following a single dose | Days 1, 5 and 19
Number and percent of subjects having a maximum QTcF, HR, PR, and QRS outside of pre-specified categories and those having a maximum ΔQTcF outside of pre-specified categories | Days 1, 5 and 19
Time of maximum observed plasma concentration (Tmax) of EFV | Days 1, 2, 19 and 20
Maximum observed plasma concentration (Cmax) of EFV | Days 1, 2, 19 and 20
Trough observed plasma concentration 24 h after a dose (C24) of EFV | Days 1, 2, 19 and 20
Area under the concentration-time curve in one dosing interval (AUC(TAU)) of EFV | Days 1, 2, 19 and 20
Safety based on incidence of AEs, SAEs, AEs leading to discontinuation, marked laboratory abnormalities, findings on 12-lead safety ECG measurements and physical examinations, and abnormalities in vital sign measurements exceeding pre-defined thresholds | Up to 30 days after discontinuation of dose (approximately 52 days)
  Serious AE (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Parexel International - Baltimore Epcu, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Abdelhady AM, Shugg T, Thong N, Lu JB, Kreutz Y, Jaynes HA, Robarge JD, Tisdale JE, Desta Z, Overholser BR. Efavirenz Inhibits the Human Ether-A-Go-Go Related Current (hERG) and Induces QT Interval Prolongation in CYP2B6*6*6 Allele Carriers. J Cardiovasc Electrophysiol. 2016 Oct;27(10):1206-1213. doi: 10.1111/jce.13032. Epub 2016 Jul 25. PMID 27333947
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx